CLINICAL TRIAL: NCT06043258
Title: Clinical and Radiographic Assessment of Bond Apatite in Horizontal Bone Augmentation Around Dental Implant
Brief Title: Bond Apatite in Horizontal Augmentation Versus Bio-Oss
Acronym: BondApatite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M07061119
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Horizontal Ridge Deficiency
MeSH Terms: interventions — Bio-Oss

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group I) study group (Experimental): eight patients with missing anterior or premolar tooth with insufficient horizontal (bucco/labio palatal) bone width were treated with dental implants and Bond Apatite (AugmaBio, United States of America) as a bone graft material to fill the defect.
  Interventions: Other: Bond Apatite
- (Group II) positive control group (Active Comparator): eight patients with missing anterior or premolar tooth with insufficient horizontal (bucco/labio palatal) bone width were treated with dental implants and Bio-Oss (Bio-Oss, GeistlichPharmaAG, Wolhusen, Switzerland) as a bone graft material to fill the defect and pericardium resorbable membrane.
  Interventions: Other: Bio-Oss

INTERVENTIONS:
Other: Bond Apatite — composite graft formed of biphasic calcium sulphate and hydroxyapatite at a ratio of 2:1
  Arms: (Group I) study group
Other: Bio-Oss — xenograft bone substitute
  Arms: (Group II) positive control group

SUMMARY:
Sixteen healthy patients selected from the Outpatient Clinic of the Department of Oral Medicine, Periodontology, Diagnosis and Oral Radiology, Faculty of Dentistry, Mansoura University for the replacement of missing single maxillary anterior or premolar tooth (in the esthetic zone) by dental implant. Patients were selected according to the following criteria: 1) Patients older than 18 years. 2) Good general health, with no systemic diseases that might contraindicate receiving a dental implant. 3) Every patient should have at least one missing tooth in the maxillary anterior premolar area and subsequently scheduled for implant supported prosthesis. 4) The tooth has been extracted from at least 3 months. 5) Insufficient horizontal bone (class III according to Len Tolstunov classification. 6) Good oral hygiene.

Patients were classified into two groups:

Group (I) (study group): eight patients with missing anterior or premolar tooth with insufficient horizontal (bucco/labio palatal) bone width were treated with dental implants and Bond Apatite (AugmaBio, United States of America) as a bone graft material to fill the defect.

Group (II) (positive control group): eight patients with missing anterior or premolar tooth with insufficient horizontal (bucco/labio palatal) bone width were treated with dental implants and Bio-Oss (Bio-Oss, GeistlichPharmaAG, Wolhusen, Switzerland) as a bone graft material to fill the defect and pericardium resorbable membrane.

Patients were evaluated with the following clinical and radiological parameters presurgical and 12 months after operation:

A) Clinical evaluation:

The following parameters were evaluated:

1. Modified plaque index:

   This is fundamentally based on the visual detection of plaque, it ascertains the thickness of plaque along the gingival margin, namely the desirability of distinguishing clearly between severity and the location of soft debris aggregates.
2. Modified gingival index:

   It is a method to assess the severity of gingivitis based on gingival color, contour, presence of bleeding, stippling and crevicular fluid flow. It is completely noninvasive method (only visual).
3. Probing depth:

Peri-implant pocket depth was measured using plastic implant probe (contrast PA probe # CPNG22, Helmut Zepf Medizintechnik Gmbh®) after final restoration was inserted.

B) Radiographic evaluation:

Bone width was assessed using CBCT 12 months after implant insertion. Bone width measurements were made on tomographic slices perpendicular to the longitudinal axis of the alveolar crest; 2 mm from the alveolar crest.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Good general health.
* Able to provide informed consent.
* Availability for multiple follow up appointments.
* Every patient should have at least one missing tooth in the maxillary anterior premolar area and subsequently scheduled for implant supported prosthesis.
* The tooth has been extracted from at least 3 months.
* Insufficient horizontal bone (class III according to Len Tolstunov classification.
* Good oral hygiene.

Exclusion Criteria:

* History of systemic disease that will contraindicate intraoral surgical procedures.
* Chronic treatment with any medication known to affect oral status and bone turnover.
* Surgical procedures within 30 days of study initiation.
* Long term nonsteroidal anti-inflammatory drugs exceeding 100 mg per day.
* Pregnant or lactating women.
* Acute dentoalveolar infection
* Smokers more than 10 cigarettes per day.
* Uncontrolled or untreated periodontal disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Bone width gain measurement | 12 months
  CBCT used to assess horizontal bone measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed Farrag, Damietta, Egypt